CLINICAL TRIAL: NCT07384676
Title: A Large-Scale Prospective Cohort Study on the Association of Environmental Exposures and Behavioral Factors With Infertility and Assisted Reproductive Technology (ART) Success Rates
Brief Title: Environmental and Behavioral Factors in Infertility and ART Outcomes
Status: Recruiting | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Peng enuo, Department Director, The Third Xiangya Hospital of Central South University
Other Study IDs: xy3-Peng-ENV
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Environmental Exposure; Assisted Reproductive Technology; Prospective Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group
  Interventions: Behavioral: plastic products
- Non-exposure group
  Interventions: Behavioral: None exposure

INTERVENTIONS:
Behavioral: plastic products — Environmental pollutants related to plastic products
  Groups: Exposure group
Behavioral: None exposure — No environmental pollutants related to plastic products
  Groups: Non-exposure group

SUMMARY:
This large-scale study aims to understand how everyday environment and lifestyle may affect the success of fertility treatments like IVF. The main idea is that exposure to certain environmental chemicals (e.g., from plastics or air pollution) and personal habits (e.g., diet, stress) could be linked to whether these treatments result in a successful pregnancy and live birth.

The study will follow approximately 5,000 couples undergoing fertility treatment in Hunan, China. Participants will answer questionnaires about their health, lifestyle, and environment and provide small biological samples (like blood and urine) during their standard treatment process. Their treatment outcomes will be tracked anonymously.The goal is to identify factors that might lower the chances of treatment success. This knowledge could help future patients and doctors make informed decisions and could guide public health advice on reducing potential risks. The study has received ethical approval, and all participant information will be kept strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* A. Women aged 18 to 46 who use their own eggs; Men aged 18 to 55 who use their own sperm; B. Patients meeting the diagnostic criteria for infertility; C. Medical history clearly indicating the duration of persistent infertility; D. Voluntarily participating in the project and signing the informed consent form;

Exclusion Criteria:

* A. The groups of artificial insemination patients with any of the following ARTs contraindications: a. The female has a sperm-egg combination disorder caused by tubal factors. b. The female has acute infections of the reproductive and urinary systems or sexually transmitted diseases. c. The female has genetic diseases, severe physical illnesses, or mental and psychological disorders. d. There is a history of giving birth to infants with congenital defects and it has been confirmed that the defect was caused by the female. e. The female has been exposed to teratogenic doses of radiation, toxins, or drugs and is in the active period. f. The female has bad habits such as alcoholism or drug abuse. B. The groups of first-generation and second-generation IVF patients with any of the following ARTs contraindications: a. Either of the parties providing gametes has acute infections of the reproductive and urinary systems and sexually transmitted diseases or has bad habits such as alcoholism or drug abuse. b. Either of the parties providing gametes has been exposed to teratogenic doses of radiation, toxins, or drugs and is in the active period. c. The female partner of the recipient who provides eggs or embryos has acute infections of the reproductive and urinary systems and sexually transmitted diseases, or has bad habits such as alcoholism or drug abuse. d. The female has an unviable uterus or severe physical illnesses that cannot withstand pregnancy. C. No embryo transfer was performed after egg retrieval; D. More than 180 days have passed since egg retrieval and frozen embryo transfer was performed.

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study aims to establish a cohort of infertility patients in Hunan Province. Patients with infertility who visited Xiangya Third Hospital in Changsha, Hunan Province from December 2024 to December 2034 will be included. The research subjects will be selected based on clear inclusion and exclusion criteria. Baseline data covering social demographic characteristics, lifestyle behaviors, basic health status, physiological and biochemical indicators, and exposure measurements of environmental factors will be collected from the start of the study to follow-up until the time of childbirth, pregnancy, delivery, and postpartum care, to observe the live birth situation of infertility patients through ART. This will provide data support for the research on identifying risk factors, early prediction, intervention and prevention of infertility patients' ART.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate following the first ART cycle | Within 24 months from the initiation of the first ART cycle
  The proportion of participants achieving at least one live birth (gestational age ≥ 28 weeks) after the initiation of their first ART treatment cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center of Xiangya Third Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT07384676/Prot_SAP_000.pdf